CLINICAL TRIAL: NCT00554489
Title: A Feasibility Study of a Physical Activity Intervention in Older Adult Inpatients With Acute Leukemia
Brief Title: Physical Activity in Older Patients With Acute Myeloid Leukemia Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000573938; CCCWFU-98107; IRB00003355
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: exercise intervention — participation in physical activity intervention program weeks 2 through 5

SUMMARY:
RATIONALE: Physical activity sessions may help improve physical function, quality of life, and symptoms caused by chemotherapy in older patients with acute myelogenous leukemia.

PURPOSE: This clinical trial is studying how well physical activity works in improving quality of life in older patients with acute myelogenous leukemia undergoing chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To test the feasibility of conducting a physical activity intervention in hospitalized older adults with acute myeloid leukemia (AML) undergoing induction or reinduction chemotherapy.

Secondary

* To obtain preliminary data regarding the effectiveness of a physical activity intervention on physical function, quality of life, and treatment-related symptoms in these patients.

OUTLINE: Patients undergo a baseline evaluation in week 1 focusing on basic demographics, health, physical function and quality-of-life assessments. These assessments include the Short Physical Performance Battery (SPPB); the Hand Grip Test of Muscular Strength; the Demographics and Physical Activity History; the Functional Assessment of Cancer Therapy (FACT-Leu); the Distress Thermometer; the Short-form Positive Affect Schedule (PANAS-SF); the Satisfaction with Life Scale (SWL); the FAST-23 Disability Measure; the Center for Epidemiologic Studies Depression Scale Short Form (CES-D); the Self-efficacy for Physical Activity Scale; the Intervention Feedback Form; and the Pre-Post Session Ratings. Some medical data may be obtained from the patient's medical record to assist in these assessments.

Beginning in weeks 2-5, patients undergo a 30-minute orientation to the exercise sessions that will be tailored to individual needs and abilities. Patients undergo a 30- to 45-minute group physical activity session twice a week, and a supervised individual session following the same format as the group session, once a week for 4 weeks. After completion of the physical activity intervention, patients complete an activities packet and repeat the physical function and quality of life assessments in weeks 5-6 and again upon readmission for consolidation therapy in weeks 9-13 .

After completion of study intervention, patients are followed for 4 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute myeloid leukemia (AML) by WHO criteria
* Planning to undergo induction or reinduction chemotherapy
* Inpatient status at Wake Forest University Baptist Medical Center
* Must not require intensive care unit support

PATIENT CHARACTERISTICS:

* Able to understand English
* Medical eligibility confirmed with Leukemia Service Attending
* Ambulatory or able to walk with a cane
* No hemodynamic instability
* No acute thrombosis within the past 7 days
* No active ischemia within the past 7 days
* No uncontrolled pain
* Must have < 3 incorrect responses on the Pfeiffer Mental Status Exam

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-07; Primary Completion 2008-11 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Percentage of adults 50 years of age or older admitted for induction or reinduction chemotherapy for acute myeloid leukemia (AML) who are eligible for the study | day 1
Percentage of eligible patients recruited into the study | day 1
Number and frequency of reported barriers to eligibility and enrollment | day 1
Percentage of study participants who successfully completed the physical and the psychosocial measures | week 13
Record barriers to completion of the physical activity program | week 13

SECONDARY OUTCOMES:
Physical function as measured by the Short Physical Performance Battery (SPPB) | week 13
Quality of Life as measured with the Distress Thermometer | week 13

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne C. Danhauer, PhD, Study Chair — Wake Forest University Health Sciences; Heidi D. Klepin, MD, Principal Investigator — Wake Forest University Health Sciences; Shannon Mihalko, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States